CLINICAL TRIAL: NCT06368180
Title: The Efficacy of a Robotic-assisted Gait Training in Comparison to Body Weight Supported Treadmill Training on Spatio-temporal Gait Parameters Among Ambulatory Children With Cerebral Palsy
Brief Title: The Efficacy of a RAGT & BWSTT on Children With CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Jaber Mohammed Ali Fagehi, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 439106274
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Palsy
Keywords: Children; Cerebral palsy; Robotic-assisted gait training; Body weight-supported treadmill training; Spatio-temporal gait parameters
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Robotic-assisted gait training Body weight-supported treadmill training
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic assisted gait training group (Experimental): This group had gait training using a robotic treadmill training system that uses body weight support belt, and driven gait orthoses (pediatric orthoses) for both legs.
  Interventions: Device: Robotic assisted gait training
- Body weight support treadmill training group (Active Comparator): This group had gait training using while the participant's body weight was supported over the treadmill by the Biodex Unweighting System.
  Interventions: Device: Body weight supported treadmill training

INTERVENTIONS:
Device: Robotic assisted gait training — is a robotic treadmill training system that uses body weight support to suspend patients by attaching their legs to robotic legs that help them walk
  Arms: Robotic assisted gait training group
Device: Body weight supported treadmill training — The Biodex Unweighting System was used to support the child's body weight, by an adjustable harness placed, over the treadmill.
  Arms: Body weight support treadmill training group

SUMMARY:
This study compared the effects of Robotic-assisted Gait Training (RAGT) and body weight support treadmill training (BWSTT) on spatio-temporal gait parameters and walking capacity among ambulatory children with bilateral Cerebral Palsy (CP)

DETAILED DESCRIPTION:
Demographic data were collected from patient medical records in the physiotherapy clinic at King Abdullah Specialist Children's Hospital and by completing the screening sheet . There were two intervention groups in this study. The first group received Robotic-assisted Gait Training (RAGT), while the second group received body weight support treadmill training (BWSTT). All participants from both intervention groups performed the home exercise program. All participants received 24 sessions three times per week over 8 weeks. Some participants were absent from some treatment sessions, either because they were suffering from flu, for reasons related to school, or other reasons. These participants were compensated with other sessions. Outcome measurements were assessed by a physiotherapist blinded to the group allocations. A physiotherapist assessed the participants at baseline and after treatment (at the end of 8 weeks)

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 5 to 14 years with bilateral spastic Cerebral palsy (CP) diagnosed by a pediatrician.
* Gross Motor Function Classifications (GMFCS); levels I (walks without limitation), II (walks with limitation), and III (walks using assistive devices).
* Able to follow instructions and accurately signal pain and discomfort.
* Hip and knee passive Range of Motion (ROM) within the minimum range requirement for Robotic-assisted Gait Training (RAGT) (≤ 10⁰ for hip and knee flexion contracture and ≤ 40⁰ for knee valgus).

Exclusion Criteria:

* Botox injection for lower limb within the past 4 to 6 months.
* Surgical intervention for lower limbs within an 8-month period before the examination date, including tendon release and muscle lengthening in a 1-year period prior to bone surgery.
* Children using an active drug for resisting epilepsy.
* Anatomical leg length difference greater than 2 centimeters (due to the limitations of the RAGT system).
* Bone-articular instability (joint dislocation).
* Fixed joint contractures (bone and joint deformity).
* Baclofen therapy with the use of an implanted infusion pump.
* Inhibited cast for a lower limb within 6 months of the study.
* Significant amblyopia and hearing loss.
* Skin inflammation and open skin lesion around the limb or trunk.
* Significant impairments in endurance due to a limitation in the cardiovascular system based on the patient's history.
* Maximum child weight is 135 kilograms and maximum height is 2.0 meters.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-08-30 (Actual); Primary Completion 2021-02-21 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Gait spatio-temporal parameters | 1 minute
  The Zebris gait analysis system was used in this study to obtain gait spatio-temporal parameters in children with CP. The Zebris gait analysis system consists of a platform that has a sensing area of 200 × 60 cm.

SECONDARY OUTCOMES:
Six-minute walk test (6MWT) | 6 minutes
  The 6MWT is a standardized walking test used to assess walking capacity in ambulatory children with CP. It is valid and reliable for children and adolescents who have CP and are healthy

CONTACTS AND LOCATIONS:
Overall Officials: Adel A Alhusaini, professor, Principal Investigator — Department of Rehabilitation Sciences, College of Applied Medical Sciences, King Saud University
Locations (1):
- King Abdu Aziz Medical City, Riyadh, Saudi Arabia